CLINICAL TRIAL: NCT03635775
Title: Effects of Single-session Transcranial Direct Current Stimulation in Children With Cerebral Palsy
Brief Title: Single-session tDCS in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00002820; P2CHD086844 (NIH); K01HD078484 (NIH)
Record Dates: First submitted 2018-07-12; First posted 2018-08-17 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy; Perinatal Stroke; Periventricular Leukomalacia
Keywords: non-invasive brain stimulation; rehabilitation; pediatrics
MeSH Terms: conditions — Cerebral Palsy; Leukomalacia, Periventricular | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and families will be masked to intervention group. The research team members performing assessments will be masked to intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Anodal ipsilesional Active tDCS (Experimental): Anodal tDCS (excitatory) applied to the lesioned hemisphere. Participant must have lesioned hemisphere MEP.
  Interventions: Device: Active tDCS
- Cathodal contralesional Active tDCS (Experimental): Cathodal tDCS (inhibitory) applied to the non-lesioned hemisphere. Participant must have lesioned hemisphere MEP.
  Interventions: Device: Active tDCS
- Anodal contralesional Active tDCS (Experimental): Anodal tDCS (excitatory) applied to the non-lesioned hemisphere. Participant must not have lesioned hemisphere MEP.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Sham tDCS applied in one of the above configurations
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Low-level (1.5 milliampere) current delivered to the scalp using saline-soaked sponges.
  Other Names: transcranial direct current stimulation
  Arms: Anodal contralesional Active tDCS; Anodal ipsilesional Active tDCS; Cathodal contralesional Active tDCS
Device: Sham tDCS — Sham-setting--no electrical current delivered.
  Arms: Sham tDCS

SUMMARY:
The goal of this study is to characterize individual responses to a single application of transcranial direct current stimulation (tDCS) in children with unilateral cerebral palsy (UCP), and to test which electrode configuration produces changes in brain excitability and motor function. Participants with UCP, ages 7-21 years, will be assigned to one of four tDCS groups. Using single-pulse transcranial magnetic stimulation, the investigators will assess cortical excitability before and at regular intervals up to 1 hour following tDCS. The knowledge gained from this study will advance the field through more targeted approaches of neuromodulatory techniques in this population and others, using individual characteristics to guide optimal treatment

DETAILED DESCRIPTION:
Hemiparesis, or weakness on one side of the body, is common following stroke early in life. The broader clinical diagnosis for this type of childhood movement impairment is unilateral cerebral palsy (UCP). Cerebral palsy effects about 3 out of every 1000 live births in the Unites States, and produces lifelong motor, sensory, and cognitive disability.

Neurorehabilitation has primarily focused on intensive motor training to encourage use of the affected extremities in an effort to produce use-dependent neuroplasticity in the brain. Such interventions are effective, but require a burdensome amount of time, 60-90 hours per week, for both the child and therapist. Furthermore, some children do not respond at all to such training.

Neuromodulation is a relatively new field that aims to influence the brain's neuronal activity through direct application of magnetic (TMS) or electric (tDCS) energy. It is thought the combination of neuromodulation and motor training may reduce the dosage of training needed, and would promote recovery to a greater extent for more individuals. Indeed, previous work in adult stroke demonstrate a benefit of combining repetitive TMS (rTMS) and tDCS with motor training, compared to training alone. These types of synergistic interventions are just beginning to be used in children with UCP, with some preliminary data showing potential benefit.

One of the many questions surrounding neuromodulatory interventions like tDCS is how to reliably predict changes in neuronal activity. The currently hypothesized effects of tDCS are polarity-specific: anodal tDCS depolarizes membranes resulting in increased in neuronal excitability; cathodal tDCS hyperpolarizes tDCS resulting in decreased neuronal excitability. Furthermore, these effects scale with the intensity of stimulation: the larger the direct current delivered, the greater the change in excitability. This framework has been used to guide almost all studies using tDCS to produce a change in brain function and resulting behavior.

More recently, the field is beginning to appreciate that this framework may be overly simplistic. For example, when a cognitive task is performed concurrently with tDCS, there are reported non-linear effects related to current intensity and direction of change in excitability. Such work has a significant impact on the use of tDCS in rehabilitation, which advocates for the pairing of stimulation with on-going activity.

One common approach to using tDCS in individuals with stroke is to target the non-lesioned hemisphere. Following stroke, there is an imbalance of communication between brain hemispheres. This communication, known as interhemispheric inhibition (IHI), is a normal control process whereby the activated motor cortex sends an inhibitory command to the opposite motor cortex to momentarily interrupt its activity, allowing for the execution of controlled unilateral movements. IHI is exaggerated in the non-lesioned hemisphere after stroke, resulting in increased inhibition on the lesioned hemisphere. Applying inhibitory current to the non-lesioned hemisphere may disinhibit this side and allow for recovery in the lesioned hemisphere.

IHI is mediated through fibers passing through the corpus callosum and can be examined non-invasively using TMS. First and foremost, IHI has been shown to exist in children and young adults, indicating that this mechanism is not exclusively a feature of the developed adult nervous system. The effect of NIBS to modulated IHI has been demonstrated in adults with stroke, but less clearly in children. One reason for this is a lack of data characterizing IHI in children after perinatal brain injury. It is feasible, through ongoing adaptive and maladaptive neuroplasticity, that IHI is weakly present (or not at all) in these children as compared to adults. As studies continue to focus on NIBS interventions targeting the non-lesioned hemisphere, a more comprehensive understanding of the motor control mechanisms present in children with UCP is needed to guide these interventions. Therefore, one objective of this study is to characterize IHI of both brain hemispheres in children with UCP.

At the moment, it is unclear what the acute effects of a single session tDCS are, when paired with motor training, on brain excitability or motor performance in children with and without UCP. This leads this investigative team to design the proposed study, which will offer insight into the mechanisms of tDCS and lead the field toward a better understanding of how tDCS be implemented in a neurorehabilitation setting for both children and potentially adults.

Purpose: To characterize motor cortex neurophysiology and to understand how one form of non-invasive brain stimulation (NIBS) called transcranial direct current stimulation (tDCS) changes brain excitability and behavior in children diagnosed with cerebral palsy, as compared to children with typical development (CTD).

Aim 1: Using transcranial magnetic stimulation (TMS), characterize brain excitability, specifically interhemispheric inhibition, in children with CP and CTD.

Aim 2: Evaluate the immediate effect of tDCS on brain excitability and motor performance in children with UCP and CTD.

Aim 3: Compare the responses to tDCS in each with individual estimated electric field intensity from computational modeling.

Procedures:

This is a randomized, sham-controlled, double-blinded study. The intervention consists of a single, 20 minute session of tDCS paired with motor training (see Figure 2). Participants will be randomized to either real or sham tDCS. The participants and the members of the research team involved in assessments and testing will be blinded to intervention group (real or sham tDCS), but the other research staff/PI/Co-Is will be unblinded.

The investigators will complete TMS assessments of cortical excitability at Pre-test, as well as an MRI of the brain. Behavioral assessments of hand function and performance will also be included.

The intervention will last a total of 30 minutes, including preparatory time. Participants will be randomly assigned to receive real or sham tDCS. Children with presence of a lesioned hemisphere motor evoked potential (MEP) response may receive 1) ipsilesional anodal; 2) contralesional cathodal tDCS or 3) sham tDCS. Children without a lesioned hemisphere MEP may receive 1) contralesional anodal or 2) sham tDCS. Participants and their families will be blinded to group assignment. Participants will be unblinded after completing the study.

Immediately following the intervention, TMS and Behavioral assessments will be performed at 0, 15, 30, and 60 minutes following the intervention.

Study Duration: Each participant will complete the study in either one day (MRI and intervention, four hours total) or on two separate days (one hour MRI, and three hours intervention). If done on two days, the MRI and intervention will be separated by no longer than a two week (14 day) period.

ELIGIBILITY:
Inclusion Criteria (for all participants):

* Ages 7-21
* Able to follow two-step commands.
* Presence of an MEP in the non-lesioned hemisphere

Exclusion Criteria (for all participants):

* Evidence of seizure within 2 years
* Other neurological or metabolic conditions
* Is pregnant (females only)
* Presence of indwelling metal in the head (e.g. aneurysm clip) or medical device.

Inclusion Criteria (for participants with cerebral palsy):

* Clinical diagnosis of unilateral cerebral palsy
* Radiological evidence of stroke or periventricular leukomalacia

Exclusion Criteria(for participants with cerebral palsy):

* Treatment with injectable agents (e.g. Botox) for spasticity management within 2 months

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samuel Nemanich, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen D, Van Naarden Braun K, Doernberg NS, Maenner MJ, Arneson CL, Durkin MS, Benedict RE, Kirby RS, Wingate MS, Fitzgerald R, Yeargin-Allsopp M. Prevalence of cerebral palsy, co-occurring autism spectrum disorders, and motor functioning - Autism and Developmental Disabilities Monitoring Network, USA, 2008. Dev Med Child Neurol. 2014 Jan;56(1):59-65. doi: 10.1111/dmcn.12268. Epub 2013 Oct 1. PMID 24117446
- [Background] Bolognini N, Vallar G, Casati C, Latif LA, El-Nazer R, Williams J, Banco E, Macea DD, Tesio L, Chessa C, Fregni F. Neurophysiological and behavioral effects of tDCS combined with constraint-induced movement therapy in poststroke patients. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):819-29. doi: 10.1177/1545968311411056. Epub 2011 Jul 29. PMID 21803933
- [Background] Figlewski K, Blicher JU, Mortensen J, Severinsen KE, Nielsen JF, Andersen H. Transcranial Direct Current Stimulation Potentiates Improvements in Functional Ability in Patients With Chronic Stroke Receiving Constraint-Induced Movement Therapy. Stroke. 2017 Jan;48(1):229-232. doi: 10.1161/STROKEAHA.116.014988. Epub 2016 Nov 29. PMID 27899754
- [Background] Antal A, Terney D, Poreisz C, Paulus W. Towards unravelling task-related modulations of neuroplastic changes induced in the human motor cortex. Eur J Neurosci. 2007 Nov;26(9):2687-91. doi: 10.1111/j.1460-9568.2007.05896.x. Epub 2007 Oct 26. PMID 17970738
- [Background] Duque J, Hummel F, Celnik P, Murase N, Mazzocchio R, Cohen LG. Transcallosal inhibition in chronic subcortical stroke. Neuroimage. 2005 Dec;28(4):940-6. doi: 10.1016/j.neuroimage.2005.06.033. Epub 2005 Aug 9. PMID 16084737
- [Background] Murase N, Duque J, Mazzocchio R, Cohen LG. Influence of interhemispheric interactions on motor function in chronic stroke. Ann Neurol. 2004 Mar;55(3):400-9. doi: 10.1002/ana.10848. PMID 14991818
- [Background] Zewdie E, Damji O, Ciechanski P, Seeger T, Kirton A. Contralesional Corticomotor Neurophysiology in Hemiparetic Children With Perinatal Stroke. Neurorehabil Neural Repair. 2017 Mar;31(3):261-271. doi: 10.1177/1545968316680485. Epub 2016 Nov 24. PMID 27885162
- [Background] Kirton A, Deveber G, Gunraj C, Chen R. Cortical excitability and interhemispheric inhibition after subcortical pediatric stroke: plastic organization and effects of rTMS. Clin Neurophysiol. 2010 Nov;121(11):1922-9. doi: 10.1016/j.clinph.2010.04.021. PMID 20537584
- [Background] Collange Grecco LA, de Almeida Carvalho Duarte N, Mendonca ME, Galli M, Fregni F, Oliveira CS. Effects of anodal transcranial direct current stimulation combined with virtual reality for improving gait in children with spastic diparetic cerebral palsy: a pilot, randomized, controlled, double-blind, clinical trial. Clin Rehabil. 2015 Dec;29(12):1212-23. doi: 10.1177/0269215514566997. Epub 2015 Jan 20. PMID 25604912
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Gillick BT, Krach LE, Feyma T, Rich TL, Moberg K, Thomas W, Cassidy JM, Menk J, Carey JR. Primed low-frequency repetitive transcranial magnetic stimulation and constraint-induced movement therapy in pediatric hemiparesis: a randomized controlled trial. Dev Med Child Neurol. 2014 Jan;56(1):44-52. doi: 10.1111/dmcn.12243. Epub 2013 Aug 21. PMID 23962321
- [Background] Kirton A, Chen R, Friefeld S, Gunraj C, Pontigon AM, Deveber G. Contralesional repetitive transcranial magnetic stimulation for chronic hemiparesis in subcortical paediatric stroke: a randomised trial. Lancet Neurol. 2008 Jun;7(6):507-13. doi: 10.1016/S1474-4422(08)70096-6. Epub 2008 May 1. PMID 18455961
- [Background] Ciechanski P, Kirton A. Transcranial Direct-Current Stimulation Can Enhance Motor Learning in Children. Cereb Cortex. 2017 May 1;27(5):2758-2767. doi: 10.1093/cercor/bhw114. PMID 27166171
- [Background] Kirton A, Ciechanski P, Zewdie E, Andersen J, Nettel-Aguirre A, Carlson H, Carsolio L, Herrero M, Quigley J, Mineyko A, Hodge J, Hill M. Transcranial direct current stimulation for children with perinatal stroke and hemiparesis. Neurology. 2017 Jan 17;88(3):259-267. doi: 10.1212/WNL.0000000000003518. Epub 2016 Dec 7. PMID 27927938
- [Background] Bikson M, Grossman P, Zannou AL, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Response to letter to the editor: Safety of transcranial direct current stimulation: Evidence based update 2016. Brain Stimul. 2017 Sep-Oct;10(5):986-987. doi: 10.1016/j.brs.2017.06.007. Epub 2017 Jul 12. No abstract available. PMID 28734680
- [Background] Giacobbe V, Krebs HI, Volpe BT, Pascual-Leone A, Rykman A, Zeiarati G, Fregni F, Dipietro L, Thickbroom GW, Edwards DJ. Transcranial direct current stimulation (tDCS) and robotic practice in chronic stroke: the dimension of timing. NeuroRehabilitation. 2013;33(1):49-56. doi: 10.3233/NRE-130927. PMID 23949028
- [Background] Lazzari RD, Politti F, Santos CA, Dumont AJ, Rezende FL, Grecco LA, Braun Ferreira LA, Oliveira CS. Effect of a single session of transcranial direct-current stimulation combined with virtual reality training on the balance of children with cerebral palsy: a randomized, controlled, double-blind trial. J Phys Ther Sci. 2015 Mar;27(3):763-8. doi: 10.1589/jpts.27.763. Epub 2015 Mar 31. PMID 25931726
- [Background] Gillick BT, Feyma T, Menk J, Usset M, Vaith A, Wood TJ, Worthington R, Krach LE. Safety and feasibility of transcranial direct current stimulation in pediatric hemiparesis: randomized controlled preliminary study. Phys Ther. 2015 Mar;95(3):337-49. doi: 10.2522/ptj.20130565. Epub 2014 Nov 20. PMID 25413621
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Background] Gillick B, Rich T, Nemanich S, Chen CY, Menk J, Mueller B, Chen M, Ward M, Meekins G, Feyma T, Krach L, Rudser K. Transcranial direct current stimulation and constraint-induced therapy in cerebral palsy: A randomized, blinded, sham-controlled clinical trial. Eur J Paediatr Neurol. 2018 May;22(3):358-368. doi: 10.1016/j.ejpn.2018.02.001. Epub 2018 Feb 11. PMID 29456128

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anodal Ipsilesional Active tDCS | Cathodal Contralesional Active tDCS | Anodal Contralesional Active tDCS | Sham tDCS
Started | 5 | 0 | 5 | 10
Completed | 5 | 0 | 5 | 9
Not Completed | 0 | 0 | 0 | 1
Not completed — Did not meet final inclusion criteria based on initial evaluation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who completed baseline testing are included in the baseline characteristics anaylsis
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal Ipsilesional Active tDCS | Cathodal Contralesional Active tDCS | Anodal Contralesional Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 5 | 0 | 5 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 0 | 3 | 9 | 17
  Between 18 and 65 years | 0 | 0 | 2 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 6 | 10
  Male | 2 | 0 | 4 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 0 | 4 | 8 | 17
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Evoked Potential Amplitude
Description: Motor evoked potential is a measure of cortical excitability using transcranial magnetic stimulation. MEP is measured as the amplitude of electrical activity from finger muscles. Outcome is reported as the percent change in MEP amplitude from pre-intervention to immediately post-intervention.
Time Frame: approximately 5 minutes
Population: All participants for whom interventional data was collected are included in outcome measure analysis.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Anodal Ipsilesional Active tDCS | Cathodal Contralesional Active tDCS | Anodal Contralesional Active tDCS | Sham tDCS
Number analyzed (Participants) | 5 | 0 | 5 | 9
percent change | 12.4 [-102.9 to 127.8] |  | 81.7 [-39.7 to 203.1] | -34.4 [-41.5 to -26.8]

2. Secondary Outcome: Change in Movement Accuracy
Description: Finger tracking was measured using an instrumented goniometer that recorded finger position, which was then used to control a cursor on a laptop computer. The outcome is reported as the percent change in accuracy from pre-intervention to 60 minutes post-intervention.
Time Frame: Approximately 1 hours
Population: All participants for whom interventional data was collected are included in outcome measure analysis.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Anodal Ipsilesional Active tDCS | Cathodal Contralesional Active tDCS | Anodal Contralesional Active tDCS | Sham tDCS
Number analyzed (Participants) | 5 | 0 | 5 | 8
percent change | -5.67 [-69.6 to 58.2] |  | -40 [-56 to -24.1] | -28.2 [-44.6 to -11.7]

ADVERSE EVENTS:
Time Frame: Participants were monitored during the study and one day after the end of the study (follow up phone call) - approximately 2 days.
Description: No events are reported for the Cathodal Contralesional Active tCDS group, as there were no participants randomized to this condition.
Arm/Group | Anodal Ipsilesional Active tDCS | Cathodal Contralesional Active tDCS | Anodal Contralesional Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0 | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 4/5 | 0/0 | 5/5 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anodal Ipsilesional Active tDCS (N=5) | Cathodal Contralesional Active tDCS (N=0) | Anodal Contralesional Active tDCS (N=5) | Sham tDCS (N=9)
Itchiness, tingling, unusual feeling on scalp (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Tiredness/Sleepiness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache/pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle twiching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03635775/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03635775/Prot_SAP_001.pdf